CLINICAL TRIAL: NCT01230021
Title: A Phase 3b Trial Investigating the Pharmacokinetics and Safety Profile of a Single Intravenous Dose of rFXIII in Paediatric (1 to Less Than 6 Years Old) Subjects With Congenital FXIII A-subunit Deficiency
Brief Title: Safety of a Single Intravenous Dose of Recombinant Factor XIII in Children With Congenital FXIII A-subunit Deficiency
Acronym: mentor™4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F13CD-3760; U1111-1116-2533 (Other: WHO); 2009-016869-28 (EudraCT Number)
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- recombinant factor XIII (Experimental)
  Interventions: Drug: catridecacog

INTERVENTIONS:
Drug: catridecacog — Intravenous injection of a single dose of recombinant factor XIII, 35 IU/kg bodyweight

SUMMARY:
This trial is conducted in Europe and United States of America (USA). The aim of this clinical trial is to investigate the pharmacokinetics (at which rate the substance is distributed and eliminated from the body) and the safety profile of catridecacog (recombinant factor XIII (rFXIII)) in children with congenital FXIII A-subunit deficiency. Young children (1 to less than 6 years old) with congenital FXIII deficiency are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent by subject's parents or subject's legally acceptable representative before any trial related activities. Trial related activities are any procedures that would not have been performed during the normal management of the subject
* Age 1 to less than 6 years old at the time of enrolment
* Congenital FXIII subunit-A deficiency previously documented by genotyping or evaluated by genotyping through blood sampling at screening visit
* Body weight at least 10 kg

Exclusion Criteria:

* Known antibodies to FXIII
* Hereditary or acquired coagulation disorder other than FXIII A-subunit congenital deficiency
* Platelet count (thrombocytes) of less than 50 × 10^9/L (at screening visit)
* Previous history of autoimmune disorder involving autoantibodies e.g., systemic lupus erythematosus
* Previous history of arterial or venous thromboembolic events e.g., cerebrovascular accident or deep vein thrombosis
* Known or suspected allergy to trial product or related products
* Any surgical procedure in the 30 days prior to enrolment and any planned surgery during the trial period
* Any disease or condition which, judged by the Investigator, could imply a potential hazard to the subject or interfere with the trial participation or trial outcome including renal and/or liver dysfunction

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (10):
- United States (4):
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Columbus, Ohio
- Novo Nordisk Investigational Site, Petah Tikva, Israel
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Birmingham
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Newcastle upon Tyne
  - Novo Nordisk Investigational Site, Reading

REFERENCES:
- [Result] Williams M, Will A, Stenmo C, Rosholm A, Tehranchi R. Pharmacokinetics of recombinant factor XIII in young children with congenital FXIII deficiency and comparison with older patients. Haemophilia. 2014 Jan;20(1):99-105. doi: 10.1111/hae.12224. Epub 2013 Jul 9. PMID 23834599
- [Result] Brand-Staufer B, Carcao M, Kerlin BA, Will A, Williams M, Tornoe CW, Sandberg Lundblad M, Nugent D. Pharmacokinetic characterization of recombinant factor XIII (FXIII)-A2 across age groups in patients with FXIII A-subunit congenital deficiency. Haemophilia. 2015 May;21(3):380-385. doi: 10.1111/hae.12616. Epub 2015 Jan 21. PMID 25643920
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at five sites located in the UK (2 sites), Israel (1 site) and the US (2 sites).
Pre-assignment Details: Between screening and treatment with trial drug the children were assessed for eligibility. If eligible, the children were treated with one single dose of FXIII. The trial was not randomised.
Groups:
- Recombinant Factor XIII: One single dose of 35 IU/kg rFXIII was administered as an intravenous (i.v.) injection to each child. The trial included one screening visit, one treatment visit (including pharmacokinetics (PK) assessments up to 24 hours) and 4 follow-up visits (at 7, 14, 21 and 30 days after dosing). Blood samples for PK assessments were drawn pre-dose and up to 30 days after dosing.
Period: Overall Study
Arm/Group | Recombinant Factor XIII
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.67 (1.03)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration vs. Time Curve (AUC)
Description: A measure of the exposure. Blood samples for the PK assessment were drawn pre-dose and up to 30 days after dosing. The PK of FXIII in children was assessed after a single i.v. dose of rFXIII 35 IU/kg.
Time Frame: At pre-dose, 30 minutes, 24 hours, 7, 14, 21 and 30 days after dosing
Population: The full analysis set including all 6 children exposed to FXIII. All 6 children were exposed to one dose of trial product.
Measure: Mean (Standard Deviation); unit: IU*h/mL
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
IU*h/mL | 250.25 (31.19)

2. Secondary Outcome: Area Under the Concentration vs. Time Curve (AUC0-∞)
Description: A measure of exposure.
Time Frame: From day 0 to day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU*h/mL
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
IU*h/mL | 403.18 (92.20)

3. Secondary Outcome: Maximum Plasma Concentration (Cmax) for FXIII
Description: Maximum plasma concentration of the drug reached.
Time Frame: At pre-dose, 30 minutes, 24 hours, 7, 14, 21 and 30 days after dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
U/mL | 0.69 (0.14)

4. Secondary Outcome: Terminal Half-life (t½)
Description: Time point when half of the maximum plasma concentration is reached.
Time Frame: From day 0 to day 30
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
hours | 378 [236 to 596]

5. Secondary Outcome: Mean Residence Time (MRT)
Description: The mean residence time (MRT) of a drug in the body and related functions are derived for drugs which are intravenously administered.
Time Frame: From day 0 to day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
hours | 729.01 (265.98)

6. Secondary Outcome: Total Plasma Clearance (CL)
Description: The total plasma clearance is a measure of the elimination of a drug from the body. Drugs are excreted primarily by the kidneys into the urine. Clearance is calculated as 'CL=Dose / AUC0-30 days').
Time Frame: From day 0 to day 30
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/h/kg
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
mL/h/kg | 0.10 (0.02)

7. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Description: Volume of distribution at steady state (Vss) is the theoretical volume that the total amount of administered drug would have to occupy (if it were uniformly distributed), to provide the same concentration as it is in blood plasma at steady state. Steady state is achieved when all variables are constant in spite of ongoing processes.
Time Frame: At steady state
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
mL/kg | 66.07 (14.32)

8. Secondary Outcome: Percentage of Subjects With One or More Adverse Events (AEs) Recorded
Time Frame: From day 0 to day 30
Population: Safety analysis population including all 6 children exposed to FXIII. All 6 children were exposed to one dose of trial product.
Measure: Number; unit: percentage (%) of subjects
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
percentage (%) of subjects | 33.3

9. Secondary Outcome: Percentage of Subjects With One or More Serious Adverse Events (SAEs)
Time Frame: From day 0 to day 30
Population: as for outcome 8
Measure: Number; unit: percentage of subjects
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
percentage of subjects | 0

10. Secondary Outcome: Percentage of Subjects With Development of Anti-rFXIII Antibodies, Including Inhibitors (Neutralising Antibodies Against Factor XIII)
Time Frame: At screening and day 30
Population: as for outcome 8
Measure: Number; unit: percentage of subjects
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
percentage of subjects
  At screening | 50
  Day 30 | 50

11. Secondary Outcome: Coagulation Related Parameters - Fibrinogen
Time Frame: Day 0 and at day 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
g/L
  Pre-dose | 3.26 (1.04)
  Post-dose 30 days | 3.46 (0.82)

12. Secondary Outcome: Coagulation Related Parameters - Activated Partial Thromboplastin Time (aPTT, Seconds)
Time Frame: Day 0 and day 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Sec
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
Sec
  Pre-dose | 33.8 (9.0)
  Post-dose | 30.3 (5.6)

13. Secondary Outcome: Coagulation Related Parameters - Prothrombin Time (PT) (Seconds)
Time Frame: Day 0 and day 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Sec
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
Sec
  Pre-dose | 12.6 (0.7)
  Post-dose | 12.1 (2.3)

14. Secondary Outcome: Clot Solubility Test (Evaluated as Normal/Abnormal)
Description: Blood samples for clot solubility drawn at each visit (1 hour before and after dose administration). A clot solubility assay was used to screen for FXIII deficiency. The assay is based on the ability of urea to dissolve fibrin clots that have not undergone FXIII-induced stabilization. Normal blood clots generally remain stable for 24 hours or more, while clots in which fibrin molecules have not been cross-linked are soluble within minutes. The outcome of the test is normal (FXIII present; a clot is observed in the test tube) or abnormal (FXIII absent or very low level; no clot in test tube).
Time Frame: Day 0 and day 30
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
participants
  Normal (pre-dose) | 4
  Abnormal (pre-dose) | 1
  Not done (pre-dose) | 1
  Normal (post-dose) | 5
  Abnormal (post-dose) | 0
  Not done (post-dose) | 1

15. Secondary Outcome: Vital Signs - Pulse
Time Frame: Day 0 and day 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
beats/minute
  pre-dose | 95.3 (14.3)
  post-dose | 113.2 (10.6)

16. Secondary Outcome: Vital Signs - Blood Pressure (Systolic and Diastolic)
Time Frame: Day 0 and day 30
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
mmHg
  Systolic pre-dose | 98.5 (10.9)
  Systolic post-dose | 107.0 (13.7)
  Diastolic pre-dose | 59.8 (12.1)
  Diastolic post-dose | 64.0 (7.6)

17. Secondary Outcome: Physical Examination (Evaluated as Normal/Abnormal)
Time Frame: From day 0 to day 30
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Recombinant Factor XIII
Number analyzed (Participants) | 6
participants
  Normal (pre-dose) | 6
  Abnormal (pre-dose) | 0
  Normal (post-dose) | 5
  Abnormal (post-dose) | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected and reported during the entire trial period; that is from day 0 (the treatment day) to day 30 (last follow-up visit).
Description: Safety analysis population including all 6 children exposed to FXIII. All 6 children were exposed to one dose of trial product.
Arm/Group | Recombinant Factor XIII
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Factor XIII (N=6)
Pyrexia (General disorders) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk (NN) reserves the right not to release data until after specified milestones, e.g., finalisation of clinical trial report. This includes the right not to release interim results of clinical trials, as release of such information can invalidate the trial results. At end of trial, one or more manuscripts will be prepared collaboratively between Investigator(s) and NN. NN reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.